CLINICAL TRIAL: NCT06451887
Title: Early Identification of Malignant Brain Edema in laRge Artery oCclusive Stroke After Endovascular Therapy (EMBRACE Study)
Acronym: EMBRACE
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024058
Record Dates: First submitted 2024-05-27; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Endovascular Therapy; Brain Edema; Prediction Model; Ischemic Stroke
Keywords: Endovascular therapy; Brain edema; Prediction model; Ischemic stroke
MeSH Terms: conditions — Brain Edema; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To design and validate a predictive model for malignant brain edema after endovascular thrombectomy.

DETAILED DESCRIPTION:
Stroke is a significant global cause of death and disability. Endovascular thrombectomy (EVT) is currently the best treatment for acute large vessel occlusion stroke (ALVOS), as it can greatly reduce mortality and improve patient outcomes. However, only half of patients who undergo EVT achieve functional independence, and malignant brain edema (MBE), a severe complication, can occur after the procedure, leading to a poor prognosis. Previous studies have confirmed the effectiveness of early decompressive hemicraniectomy in reducing morbidity and mortality in patients with malignant brain edema. Therefore, identifying high-risk patients for MBE can help clinicians make appropriate triage and early intervention decisions, potentially saving patients' lives.

Predictive factors for post-ischemic stroke brain edema have been widely discussed, and reliable early predictive indicators have been identified, such as age, early consciousness disorders, baseline National Institutes of Health Stroke Scale (NIHSS), atrial fibrillation, hypertension, baseline blood glucose, and the level of reperfusion after EVT. Radiological factors, such as the Alberta Stroke Program Early CT Score (ASPECTS), collateral circulation rating of arteries, venous outflow status, CT perfusion core infarct volume, perfusion-based collateral status, and clot burden, are closely associated with the occurrence of MBE post-EVT. However, due to individual differences and multiple factors affecting MBE, a single factor cannot effectively predict MBE. Establishing a clinical risk prediction model can effectively identify high-risk populations for MBE at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age > 18 years old; (2)Onset of stroke to hospital admission < 24 hours; (3)Admission with a head CT scan ruling out hemorrhage; (4)Patients undergoing CT perfusion scan before treatment; (5)Confirmation of internal carotid artery (ICA) or middle cerebral artery (MCA) occlusion or tandem occlusion by Digital Subtraction Angiography (DSA) and subsequent EVT; (6)complete 3-months follow-up.

Exclusion Criteria:

* (1)Poor quality of preoperative CT perfusion imaging; (2)Posterior circulation occlusion or isolated anterior cerebral artery occlusion; (3)Presence of other severe diseases such as malignant tumors, severe organ failure, or other life-threatening conditions with an expected survival period of less than 90 days; (4)Incomplete imaging and clinical data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is a multicenter, prospective, observational clinical registry study, commenced on April 1, 2024, and is expected to end in June 2027. Participants were ALVOS patients undergoing EVT treatment in neurology departments from multiple stroke centers. The data from Zhejiang Provincial People's Hospital compose the model training cohort, while data from other centers serve as an independent external validation cohort. The protocol of the study has been approved by the human Ethics Committee of Zhejiang Provincial People's Hospital (KY2024058). All clinical investigations will be conducted according to the principles set in the Declaration of the Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The occurrence of MBE | 3 days post-EVT
  Patients developed MBE within 3 days post-EVT

SECONDARY OUTCOMES:
90 days mRS score | 90 days after EVT
  The follow-up mRS scores of enrolled patients at 90 days after EVT.
PH | 3-5 days after EVT
  Evidence of parenchymal hemorrhage (PH type) on cranial imaging at 3-5 days after EVT

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT06451887/Prot_000.pdf
  • Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT06451887/ICF_001.pdf